CLINICAL TRIAL: NCT06359158
Title: Enhancing Respiratory Auscultation Skills Among Medical Students: A Randomized Controlled Trial on the Integration of Digital Stethoscopes in Medical Education
Brief Title: Enhancing Respiratory Auscultation Skills Among Medical Students: Digital Stethoscopes in Medical Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Collaborators: Ministry of Education, Taiwan (Other Government)
Responsible Party: Principal Investigator, Frank Lin, MD, PhD, Attending Physician, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: eStethoscope for Med Student
Record Dates: First submitted 2024-03-23; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Auscultation; Breathing Sound; Asthma; Pneumonia; Pleural Effusion
Keywords: Medical Education; Auscultation Pedagogy; Digital Stethoscope; Clinical Skills Training
MeSH Terms: conditions — Respiratory Sounds; Asthma; Pneumonia; Pleural Effusion | interventions — Evaluation Studies as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital stethoscope use (Experimental): The intervention comprises a comprehensive curriculum titled "Respiratory Auscultation with Digital Stethoscopes," designed to enhance the proficiency of medical students in diagnosing respiratory disorders through auscultation. The curriculum utilizes advanced digital stethoscope technology, specifically electronic digital stethoscopes, and the Eko auscultation software platform, to facilitate the visualization and analysis of recorded breath sounds, thereby augmenting traditional auscultation training methods.
  Interventions: Device: Digital stethoscope use
- Traditional stethoscope use (No Intervention): The curriculum utilizes a traditional stethoscope.

INTERVENTIONS:
Device: Digital stethoscope use — In this interventional study, 84 medical students were randomly allocated to an intervention group utilizing a novel digital stethoscope curriculum or a control group receiving traditional instruction. The intervention leveraged digital stethoscopes, enabling visualization and analysis of recorded breath sounds. Pre- and post-assessments evaluated respiratory
  Other Names: video; Pre- and Post- test; Questionnaire on student feedback
  Arms: Digital stethoscope use

SUMMARY:
Objectives: This study aims to assess the effectiveness of a novel digital stethoscope curriculum integrated into respiratory auscultation training for medical students. It seeks to compare the auscultation proficiency gained through this innovative approach with that from traditional teaching methods, to understand the potential of digital stethoscopes in reinvigorating clinical skills training.

Methods: In a single-center, controlled, longitudinal, randomized experimental design, 84 medical students undergoing clinical clerkship rotations at Chung Shan Medical University Hospital were enrolled. Participants were randomly assigned to either the intervention group, receiving training with digital stethoscopes and the Eko auscultation software, or the control group, following a traditional curriculum. Pre- and post-intervention assessments measured auscultation skills, and student feedback on teaching quality was collected. The primary outcome was the improvement in auscultation proficiency, while secondary outcomes included student engagement and feedback on the educational approach.

Expected Results: The investigators hypothesize that the integration of digital stethoscopes into the curriculum will significantly improve the auscultation skills of medical students compared to traditional methods. Enhanced engagement and positive feedback from students are anticipated, underscoring the pedagogical value of incorporating digital health technologies in medical education.

DETAILED DESCRIPTION:
Subjects and Procedures Research Methodology The present investigation carried out at a university hospital, was a longitudinal, controlled, single-center, randomized trial with an interventional design. A total of 84 medical students who were completing their clinical clerkship rotations in the Department of Thoracic Surgery were included in the study. The participants were randomized to either the intervention group or the control group.

Intervention The participants in the intervention group were provided with the curriculum titled "Respiratory Auscultation with Digital Stethoscopes," which involved the use of electronic digital stethoscopes and the Eko auscultation software platform developed by Eko Devices in Berkeley, California, USA. The utilization of this methodology enabled the viewing and examination of documented respiratory sounds, which were then shown as phonopneumograms. The participants assigned to the control group were provided with conventional respiratory auscultation training in accordance with the established clerkship curriculum. The curriculum encompassed practical sessions conducted at the Objective Structured Clinical Examination (OSCE) center, utilizing the SAM II respiratory sound simulator (Cardionics, Webster, Texas, USA). Additionally, instructional videos were provided to facilitate the acquisition of knowledge pertaining to breath sounds. Furthermore, a breathing assignment was assigned to each student, necessitating the recording and description of five distinct breath sounds. The process of gathering data The Zuvio Interactive Response System (Zuvio, Taipei, Taiwan) was used to measure participants' auscultation skills before and after the intervention. This was done by employing a question bank consisting of 50 breath sound audio files. The collection of student feedback regarding the quality of teaching and the helpfulness of the course was conducted by means of surveys employing 5-point Likert scales. Furthermore, the researchers collected data pertaining to OSCE attendance, video viewing, answer-checking behavior, and the time interval between pre-and post-tests. The variables that were assessed included alterations in auscultation test scores and self-reported levels of teaching satisfaction within the two cohorts.

Statistical analysis The data analysis was performed utilizing the Statistical Package for Social Sciences (IBM SPSS Statistics, version 25). A range of statistical tests were employed to comprehensively analyze the distribution of student scores and teaching satisfaction, compare the intervention and control groups, and explore the influence of the course on students' engagement and learning outcomes. The normality of distributions for student scores and teaching satisfaction was initially examined using the Kolmogorov-Smirnov test. To compare scores and satisfaction levels between the intervention and control groups, either the Student t-test or the Mann-Whitney U test was selected, depending on the distributions. The paired Student's t-test or the Wilcoxon signed-rank test was used, as appropriate, to assess the changes in scores before and after the course. The study employed the chi-square test to examine the disparity in the proportions of students from both groups who opted to rent electronic stethoscopes subsequent to the completed course. This was conducted as an indirect method to assess the student's level of interest in auscultation and their comprehension of digital stethoscope technology, hence indicating the effectiveness of the course instruction. In addition, the researchers used regression analysis to investigate the relationships between different variables and outcomes, thereby offering valuable insights into the determinants that impact students' learning experiences and preferences. The statistical significance level was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

Medical students who were completing their clinical clerkship rotations in the Department of Thoracic Surgery during the study period.

Exclusion Criteria:

All medical students who did not complete the clinical clerkship rotations, the pre- and post-tests, and the course feedback questionnaire.

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Pre-test and Post-test using the Zuvio Interactive Response System (Zuvio, Taipei, Taiwan) | At the beginning and end of the two-week Thoracic Surgery clinical rotation.
  The Zuvio Interactive Response System evaluates participants' auscultation skills through a question bank of 50 breath sound audio files.
Student Feedback | End of the two-week Thoracic Surgery clinical rotation.
  Helpfulness of the course: Student feedback on teaching quality and course helpfulness was collected through surveys using 5-point Likert scales.

CONTACTS AND LOCATIONS:
Overall Officials: Frank CF Lin, MD, PhD, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, South, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided